CLINICAL TRIAL: NCT06306976
Title: Assessment of the Ability to Predict Fascial Closure Using Shear-wave Elastography in Patients With Midline Incisional Hernias.
Brief Title: Shear-Wave Elastography
Acronym: ELASTOGRAPHY
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2066031
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Ventral Incisional Hernia
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: Specific Aim 1:
  Determine the elasticity of abdominal wall muscles (rectus abdominis, external oblique, internal oblique, and transversus abdominis) through shear wave elastography in patients with midline incisional hernias of varying complexity and morphology.
  Specific Aim 2:
  Correlate shear wave elastography measurements of the abdominal wall with the extent of MFR required to achieve fascial closure.
  Specific Aim 3:
  Correlate SWE-determined elasticity of abdominal wall to intraoperative assessment of tension required to achieve fascial closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group 1 (Other): Control group 1 patients will have no incisional hernia or prior laparotomy.
  Imaging:
  Ultrasound procedure will involve the following steps:
  1. For control group 1 and group 2 patients, Images will be taken at two points
  Interventions: Procedure: Imaging: Ultrasound
- Control Group 2 (Other): Control group 2 patients will have no hernia and will be undergoing elective midline laparotomy.
  Imaging:
  Ultrasound procedure will involve the following steps:
  1. For control group 1 and group 2 patients, Images will be taken at two points .
  Hernia repair:
  All study patients will have an open retromuscular repair with/without additional lateral
  Tensiometry For all study patients, an analog spring-tensiometer will be used to assess intraoperative tension required to bring the fascia to the midline for closure.
  Interventions: Procedure: Elective Midline Laparotomy; Procedure: Imaging: Ultrasound; Other: Tensiometry

INTERVENTIONS:
Procedure: Elective Midline Laparotomy — Patients with midline ventral incisional hernia with a range of hernia morphology who plan to undergo open retromuscular VHR.
  Hernia repair:
  All study patients will have an open retromuscular repair with/without additional lateral MFR (TAR or EOR at the discretion of the operating surgeon). All repairs beginning with retrorectus dissection to the level of the linea semilunaris.
  All patients will have permanent mesh reinforcement of the abdominal wall (large-pore, midweight polypropylene). Fascia will be closed over the mesh with 0 or 2-0 polydioxanone slowly absorbable suture using a small-bite technique and a 4:1 suture length:wound length ratio.
  Arms: Control Group 2
Procedure: Imaging: Ultrasound — Ultrasound procedure will involve the following steps:
  1. For control group 1 and group 2 patients, Images will be taken at two points along the bilateral RA; at the level of the umbilicus and midway between the umbilicus and xiphoid process. Bilateral external oblique (EO), internal oblique (IO), and transversus abdominis (TA) images will be performed at the level of the anterior axillary line midway between the costal margin and iliac crest.
Other: Tensiometry — For all study patients, an analog spring-tensiometer will be used to assess intraoperative tension required to bring the fascia to the midline for closure. The tensiometer is attached to a clamp attached to the fascia at the midpoint of the hernia defect. Tension required for medialization to the midline will be performed after adhesiolysis (baseline), retrorectus dissetion, incision of the PLIO (if performed), and after completion of TAR or EOR (if performed).
  Control group 2 patients will be undergoing first time laparotomy and will have tensiometry performed.
  Arms: Control Group 2

SUMMARY:
Prospective cohort study of patients with midline ventral incisional hernia with a range of hernia morphology who plan to undergo open retromuscular VHR.

Study groups: Study groups are selected across a range of morphology and based on factors known or suspected to affect the ability to achieve fascial closure.

Control groups: The study plans to enlist 5 volunteers with no incisional hernia or prior laparotomy to establish internal baseline SWE values and interrater reliability. The study will also plan to recruit 5 patients undergoing primary laparotomy in order to correlate SWE findings with closure tension.

DETAILED DESCRIPTION:
Shear wave elastography can be used to predict abdominal wall compliance pre-operatively and can therefore be used as a tool to improve surgical outcomes.

Specific Aim 1:

Determine the elasticity of abdominal wall muscles (rectus abdominis, external oblique, internal oblique, and transversus abdominis) through shear wave elastography in patients with midline incisional hernias of varying complexity and morphology.

Specific Aim 2:

Correlate shear wave elastography measurements of the abdominal wall with the extent of MFR required to achieve fascial closure.

Specific Aim 3:

Correlate SWE-determined elasticity of abdominal wall to intraoperative assessment of tension required to achieve fascial closure.

Imaging:

Ultrasound procedure will involve the following steps:

1. For control group 1 and group 2 patients, Images will be taken at two points along the bilateral RA; at the level of the umbilicus and midway between the umbilicus and xiphoid process. Bilateral external oblique (EO), internal oblique (IO), and transversus abdominis (TA) images will be performed at the level of the anterior axillary line midway between the costal margin and iliac crest.
2. For study patients, a single point of the bilateral RA will be selected at the longitudinal mid-point of the hernia defect. Bilateral EO, IO, and TA images will be performed at the level of the anterior axillary line midway between the costal margin and iliac crest.
3. Gray-scale imaging will first determine thickness and texture of each muscle layer. Texture analysis includes use of overlying subcutaneous fat as the internal control value.
4. SWE will be performed at each location with three successive maneuvers:

   1. With minimal external pressure applied by the ultrasound probe.
   2. Manual compression applied with the ultrasound probe (maximum pressure allowable without causing patient discomfort).
   3. During Valsalva.

Hernia repair:

All study patients will have an open retromuscular repair with/without additional lateral MFR (TAR or EOR at the discretion of the operating surgeon). All repairs beginning with retrorectus dissection to the level of the linea semilunaris. When needed, additional MFR progresses as follows:

1. For posterior myofascial release (TAR):

   1. Incision of the posterior lamella of the internal oblique (PLIO) just medial the intercostal neurovascular bundles and linea semilunaris
   2. Division of the transversus abdominis muscle / aponeurosisis
   3. Lateral dissection to progressively separate the peritoneum from the transversus abdominis.
2. For anterior release (EOR):

   1. Subcutaneous flaps developed to the anterior or midaxillary line bilaterally.
   2. Division of the external oblique fascial and muscle 1cm or greater from the lateral border of the rectus sheath / linea semilunaris.
   3. Lateral dissection to progressively separate the external and internal oblique muscles.

All patients will have permanent mesh reinforcement of the abdominal wall (large-pore, midweight polypropylene). Fascia will be closed over the mesh with 0 or 2-0 polydioxanone slowly absorbable suture using a small-bite technique and a 4:1 suture length:wound length ratio.

Control group 1 patients will have no incisional hernia or prior laparotomy.

Control group 2 patients will have no hernia and will be undergoing elective midline laparotomy.

Tensiometry For all study patients, an analog spring-tensiometer will be used to assess intraoperative tension required to bring the fascia to the midline for closure. The tensiometer is attached to a clamp attached to the fascia at the midpoint of the hernia defect. Tension required for medialization to the midline will be performed after adhesiolysis (baseline), retrorectus dissetion, incision of the PLIO (if performed), and after completion of TAR or EOR (if performed).

Control group 2 patients will be undergoing first time laparotomy and will have tensiometry performed. As control group 1 is not having surgery, no tensiometry will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 y/o.
* Midline ventral / incisional hernia.
* Plan for open retromuscular incisional hernia repair.

Exclusion Criteria:

* Prior VHR with mesh.
* Isolated subxiphoid (European Hernia Society (EHS) classification M1) or suprapubic hernias (EHS classification M5)
* History of flank incisions. M1 (midline position 1) is defined as the xiphoid process down to a point 3cm below the xiphoid. M5 (midline position 5) is defined as the pubis to a point 3cm above the pubis.
* Infected / contaminated cases.
* Plan for robotic, laparoscopic, or open onlay repair, or plan for primary (non-mesh) repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Determine Elasticity of Abdominal Wall Muscles (Specific Aim 1) | Study participation ends after surgery
  Determine the elasticity of abdominal wall muscles (rectus abdominis, external oblique, internal oblique, and transversus abdominis) through shear wave elastography in patients with midline incisional hernias of varying complexity and morphology using Ultrasound measurements.
Correlate Elastography measurements with MFR (Specific Aim 2) | Study participation ends after surgery
  Correlate shear wave elastography measurements of the abdominal wall with the extent of MFR required to achieve fascial closure using Ultrasound measurements.
Correlate SWE Assessment to Tensiometer (Specific Aim 3) | Study participation ends after surgery
  Correlate SWE-determined elasticity of abdominal wall to intraoperative assessment of tension required to achieve fascial closure using Tensiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Wes Love, MD, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT06306976/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT06306976/SAP_001.pdf
  • Informed Consent Form (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT06306976/ICF_002.pdf